**Mental Health Association of Hong Kong** 

1 September 2025

Consent Form for Participation in the Effectiveness Study of the "teen Mental Health

First Aid Course" for Secondary School Students

Dear Parent/Guardian,

We sincerely invite your child to participate in a research study organized by the Mental Health Association of Hong Kong on the "teen Mental Health First Aid." Mental Health

First Aid course was originally developed in Australia in 2000 and has since been shown

to effectively improve mental health awareness, including enhancing understanding of mental illnesses, reducing stigma toward individuals with mental health conditions, and

increasing motivation to seek help.

This study focuses on secondary school students and aims to understand their

knowledge of mental illnesses, attitudes toward individuals with mental health conditions, and willingness to seek help. It also evaluates the effectiveness of the course in promoting mental health literacy among participants, with the goal of refining

and localizing the program.

Participants will be asked to complete self-administered electronic questionnaires, each taking approximately 10–15 minutes. Upon completing all questionnaires, each

student will receive a HKD \$30 cash voucher. Participation is entirely voluntary, and your child may withdraw at any time without any risk or negative consequences. All data

provided will be kept confidential, used solely for research analysis, and destroyed after

the study concludes.

For inquiries, please contact Project Manager Mr. K.S. Wong

Email: kswong@mhahk.org.hk

Phone: 2180 7908

1

| Reply Slip – Parent/Guardian Consent |
|---|
| Title of Study: |
| Effectiveness Study of the "teen Mental Health First Aid Course" for Secondary School Students |
| Student Name: |
| Class: |
| School Name: |
| $\hfill\square$ I agree to allow my child to participate in the above-mentioned study. |
| $\Box$<br>I do not agree to allow my child to participate in the above-mentioned study. |
| Parent/Guardian Name: |
| Signature: |
| Date: |